CLINICAL TRIAL: NCT07375862
Title: Investigating the Clinical Benefits and Underlying Mechanisms of Danhong Injection in Modulating Mitochondrial Homeostasis Against Sepsis-Associated Myocardial Dysfunction
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY-2025-313
Record Dates: First submitted 2026-01-22; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Sepsis-Induced Myocardial Dysfunction
MeSH Terms: interventions — danhong; Sodium Chloride

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Danhong Injection (Experimental)
  Interventions: Drug: Danhong injection
- Control group (Placebo Comparator)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Danhong injection — Danhong Injection for intravenous drip, dosage: 20 ml, diluted in 80 ml of 0.9% saline solution for intravenous drip, twice daily, for a continuous treatment period of 7 days.
  Arms: Danhong Injection
Drug: Saline — Intravenous drip of 100 ml 0.9% saline solution, twice daily, for 7 consecutive days.
  Arms: Control group

SUMMARY:
This study aims to evaluate the clinical efficacy of Danhong injection in patients with septic myocardial injury through a prospective randomized controlled trial. The study will enroll 140 patients meeting criteria for septic myocardial injury, divided into a Danhong injection group and a placebo group. Primary endpoints include changes in myocardial injury markers and improvement rates in cardiac function over 7 days, while secondary endpoints include 28-day mortality rates. This will determine whether Danhong injection possesses myocardial protective effects and provide evidence-based support for expanding its clinical indications.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who met the Sepsis-3 criteria, defined by a suspected or confirmed infection and an increase in the Sequential Organ Failure Assessment (SOFA) score of 2 points or more from baseline.
2. Patients with a diagnosis of sepsis-induced myocardial dysfunction (SIMD).

Exclusion Criteria:

1. Patients with significant primary cardiac diseases, including unstable coronary artery disease, severe cardiomyopathy, or severe valvular heart disease.
2. Exclusion criteria included long-term use of Danhong Injection or recent use of other medication with potential significant impact on cardiac function.
3. Patients with severe hepatic dysfunction (defined as Child-Pugh class C) or severe renal insufficiency (defined as creatinine clearance <30 mL/min) were excluded.
4. Patients with a known allergy to any component of Danhong Injection or a history of severe allergic diathesis were excluded.
5. Pregnant or lactating women
6. Patients with severe mental illness or inability to cooperate with the study.
7. Participation in other drug clinical trials within 3 months prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Left Ventricular Ejection Fraction | 24 hours before treatment, 3 days after treatment

SECONDARY OUTCOMES:
cardiac troponin T | Before treatment, 3 days after treatment, 7 days after treatment
28-day mortality | 28 days after enrollment

IPD SHARING:
Plan to Share IPD: Undecided